CLINICAL TRIAL: NCT00105001
Title: A Randomized Phase II Study to Determine the Most Promising Postgrafting Immunosuppression for Prevention of Acute GVHD After Unrelated Donor G-CSF Mobilized Peripheral Blood Mononuclear Cell (G-PBMC) Transplantation Using Nonmyeloablative Conditioning for Patients With Hematologic Malignancies A Multi-Center Trial
Brief Title: Tacrolimus and Mycophenolate Mofetil With or Without Sirolimus in Preventing Acute Graft-Versus-Host Disease in Patients Who Are Undergoing Donor Stem Cell Transplant for Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brenda Sandmaier, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1938.00; NCI-2010-00268 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1938.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); P01CA018029 (NIH)
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Results first posted 2015-09-15 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Previously Treated Myelodysplastic Syndrome; Refractory Chronic Lymphocytic Leukemia; Refractory Plasma Cell Myeloma; Waldenstrom Macroglobulinemia; Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With t(9;11)(p22;q23); MLLT3-MLL; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Promyelocytic Leukemia With t(15;17)(q22;q12); PML-RARA; Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); RUNX1-RUNX1T1; Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Burkitt Lymphoma; Childhood Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Childhood Diffuse Large Cell Lymphoma; Childhood Immunoblastic Lymphoma; Childhood Myelodysplastic Syndrome; Stage II Contiguous Adult Burkitt Lymphoma; Stage II Contiguous Adult Diffuse Large Cell Lymphoma; Stage II Contiguous Adult Diffuse Mixed Cell Lymphoma; Stage II Contiguous Adult Diffuse Small Cleaved Cell Lymphoma; Stage II Adult Contiguous Immunoblastic Lymphoma; Stage II Contiguous Adult Lymphoblastic Lymphoma; Stage II Grade 1 Contiguous Follicular Lymphoma; Stage II Grade 2 Contiguous Follicular Lymphoma; Stage II Grade 3 Contiguous Follicular Lymphoma; Stage II Contiguous Mantle Cell Lymphoma; Stage II Non-Contiguous Adult Burkitt Lymphoma; Stage II Non-Contiguous Adult Diffuse Large Cell Lymphoma; Stage II Non-Contiguous Adult Diffuse Mixed Cell Lymphoma; Stage II Non-Contiguous Adult Diffuse Small Cleaved Cell Lymphoma; Stage II Adult Non-Contiguous Immunoblastic Lymphoma; Stage II Non-Contiguous Adult Lymphoblastic Lymphoma; Stage II Grade 1 Non-Contiguous Follicular Lymphoma; Stage II Grade 2 Non-Contiguous Follicular Lymphoma; Stage II Grade 3 Non-Contiguous Follicular Lymphoma; Stage II Non-Contiguous Mantle Cell Lymphoma; Stage II Small Lymphocytic Lymphoma; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Burkitt Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Recurrent Childhood Hodgkin Lymphoma; Recurrent Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Secondary Myelodysplastic Syndrome; Stage I Adult Burkitt Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Mixed Cell Lymphoma; Stage I Adult Immunoblastic Lymphoma; Stage I Adult Lymphoblastic Lymphoma; Stage I Childhood Anaplastic Large Cell Lymphoma; Stage I Childhood Large Cell Lymphoma; Stage I Childhood Lymphoblastic Lymphoma; Stage I Childhood Burkitt Lymphoma; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage I Marginal Zone Lymphoma; Stage I Small Lymphocytic Lymphoma; Stage II Childhood Anaplastic Large Cell Lymphoma; Stage II Childhood Lymphoblastic Lymphoma; Stage II Childhood Burkitt Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Immunoblastic Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Childhood Anaplastic Large Cell Lymphoma; Stage III Childhood Large Cell Lymphoma; Stage III Childhood Lymphoblastic Lymphoma; Stage III Childhood Burkitt Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Immunoblastic Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Childhood Anaplastic Large Cell Lymphoma; Stage IV Childhood Large Cell Lymphoma; Stage IV Childhood Lymphoblastic Lymphoma; Stage IV Childhood Burkitt Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Large-Cell, Anaplastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — fludarabine phosphate; Whole-Body Irradiation; Peripheral Blood Stem Cell Transplantation; Tacrolimus; Mycophenolic Acid; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (MMF and tacrolimus) (Active Comparator): Patients receive tacrolimus IV or PO every 12 hours on days -3 to 180 with taper beginning on day 100 in the absence of GVHD. Patients also receive MMF PO every 8 hours on days 0-29 and then every 12 hours on days 30-96 with taper beginning on day 40 in the absence of GVHD.
  Interventions: Drug: Fludarabine Phosphate; Radiation: Total-Body Irradiation; Procedure: Peripheral Blood Stem Cell Transplantation; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Tacrolimus; Drug: Mycophenolate Mofetil
- Arm II (MMF and tacrolimus alternate schedule) (Experimental): Patients receive tacrolimus IV or PO every 12 hours on days -3 to 150 with taper beginning on day 100 in the absence of GVHD. Patients also receive MMF PO every 8 hours on days 0-29 and then every 12 hours on days 30-180 with taper beginning on day 150 in the absence of GVHD.
  Interventions: Drug: Fludarabine Phosphate; Radiation: Total-Body Irradiation; Procedure: Peripheral Blood Stem Cell Transplantation; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Tacrolimus; Drug: Mycophenolate Mofetil
- Arm III (MMF, tacrolimus, and sirolimus) (Experimental): Patients receive tacrolimus and MMF as in arm II. Patients also receive sirolimus PO once daily on days -3 to 80.
  Interventions: Drug: Fludarabine Phosphate; Radiation: Total-Body Irradiation; Procedure: Peripheral Blood Stem Cell Transplantation; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Drug: Sirolimus

INTERVENTIONS:
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; SH T 586
Radiation: Total-Body Irradiation — Undergo total-body irradiation
  Other Names: TBI; Total Body Irradiation; Whole-Body Irradiation
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic peripheral blood stem cell transplantation
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic peripheral blood stem cell transplantation
  Other Names: HSC; HSCT
Drug: Tacrolimus — Given IV or PO
  Other Names: Advagraf; FK 506
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Drug: Sirolimus — Given PO
  Other Names: AY 22989; RAPA; SILA 9268A; WY-090217
  Arms: Arm III (MMF, tacrolimus, and sirolimus)

SUMMARY:
This randomized phase II trial studies how well giving tacrolimus and mycophenolate mofetil (MMF) with or without sirolimus works in preventing acute graft-versus-host disease (GVHD) in patients undergoing donor stem cell transplant for hematologic cancer. Giving low doses of chemotherapy, such as fludarabine phosphate, and total-body-irradiation before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving MMF and tacrolimus with or without sirolimus after transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine which of 3 GVHD prophylaxis regimens results in reduction of acute grades II-IV GVHD to =< 40%.

SECONDARY OBJECTIVES:

I. Reduce the incidence of non-relapse mortality from infections and GVHD before day 200 to =< 15%.

II. Reduce the utilization of high-dose corticosteroids compared to protocols 1463, 1641, and 1668.

III. Compare survival and progression-free survival to that achieved under protocols 1463, 1641, and 1668.

OUTLINE:

CONDITIONING: All patients receive fludarabine phosphate intravenously (IV) over 30 minutes on days -4 to -2 and undergo total-body irradiation on day 0.

TRANSPLANTATION: All patients undergo allogeneic peripheral blood stem cell transplantation on day 0.

IMMUNOSUPPRESSION: Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive tacrolimus IV or orally (PO) every 12 hours on days -3 to 180 with taper beginning on day 100 in the absence of GVHD. Patients also receive MMF PO every 8 hours on days 0-29 and then every 12 hours on days 30-96 with taper beginning on day 40 in the absence of GVHD.

ARM II: Patients receive tacrolimus IV or PO every 12 hours on days -3 to 150 with taper beginning on day 100 in the absence of GVHD. Patients also receive MMF PO every 8 hours on days 0-29 and then every 12 hours on days 30-180 with taper beginning on day 150 in the absence of GVHD.

ARM III: Patients receive tacrolimus and MMF as in arm II. Patients also receive sirolimus PO once daily on days -3 to 80.

After completion of study treatment, patients are followed up at 6 months and then every year thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Ages > 50 years with hematologic malignancies treatable by unrelated hematopoietic cell transplant (HCT)
* Ages =< 50 years of age with hematologic diseases treatable by allogeneic HCT who through pre-existing medical conditions or prior therapy are considered to be at high risk for regimen related toxicity associated with a conventional transplant (> 40% risk of transplant related mortality [TRM]) (This criterion can include patients with a HCT-comorbidity index (CI) score of >= 1; transplants should be approved for these inclusion criteria by both the participating institutions' patient review committees such as the Patient Care Conference (PCC) at the Fred Hutchinson Cancer Research Center (FHCRC) and by the principal investigators at the collaborating centers)
* Patients =< 50 years of age who have received previous high-dose transplantation do not require patient review committee approvals (All children < 12 years must be discussed with the FHCRC principal investigator (PI) [Brenda Sandmaier, MD 206 6674961] prior to registration)
* Ages =< 50 years of age with chronic lymphocytic leukemia (CLL); these patients do not require patient review committee approvals
* Ages =< 50 years of age with hematologic diseases treatable by allogeneic HCT who refuse a conventional HCT (Transplants must be approved for these inclusion criteria by both the participating institutions' patient review committee such as PCC at the FHCRC and by the principal investigators at the collaborating centers)
* The following diseases will be permitted although other diagnoses can be considered if approved by PCC or the participating institutions' patient review committees and the principal investigators:

  * Aggressive non-Hodgkin lymphomas (NHL) and other histologies such as Diffuse large B cell NHL not eligible for autologous hematopoietic stem cell transplant (HSCT), not eligible for conventional myeloablative HSCT, or after failed autologous HSCT
  * Mantle Cell NHL may be treated in first complete response (CR) (Diagnostic lumbar puncture [LP] required pretransplant)
  * Low grade NHL with < 6 month duration of CR between courses of conventional therapy
  * CLL must have either

    * Failed to meet National Cancer Institute (NCI) Working Group criteria for complete or partial response after therapy with a regimen containing fludarabine phosphate (FLU) (or another nucleoside analog, e.g. Cladribine [2-CDA], pentostatin) or experience disease relapse within 12 months after completing therapy with a regimen containing FLU (or another nucleoside analog);
    * Failed FLU-CY-Rituximab (FCR) combination chemotherapy at any time point; or
    * Have "17p deletion" cytogenetic abnormality; patients should have received induction chemotherapy but could be transplanted in 1st CR
  * Hodgkin Lymphoma must have received and failed frontline therapy
  * Multiple Myeloma must have received prior chemotherapy; consolidation of chemotherapy by autografting prior to nonmyeloablative HCT is permitted
  * Acute Myeloid Leukemia (AML) must have < 5% marrow blasts at the time of transplant
  * Acute Lymphocytic Leukemia (ALL) must have < 5% marrow blasts at the time of transplant
  * Chronic Myeloid Leukemia (CML) patients will be accepted if they are beyond chronic phase (CP)1 and if they have received previous myelosuppressive chemotherapy or HCT and have < 5% marrow blasts at time of transplant
  * Myelodysplasia (MDS)/Myeloproliferative Syndrome (MPS) patients must have received previous myelosuppressive chemotherapy or HCT and have < 5% marrow blasts at time of transplant
  * Waldenstrom's Macroglobulinemia must have failed 2 courses of therapy
* DONOR: FHCRC matching allowed will be Grades 1.0 to 2.1: unrelated donors who are prospectively:

  * Matched for human leukocyte antigen (HLA)-A, B, C, DRB1 and DQB1 by high resolution typing
  * Only a single allele disparity will be allowed for HLA-A, B, or C as defined by high resolution typing
* DONOR: Donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment; this determination is based on the standard practice of the individual institution; the recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain a panel reactive antibody (PRA) screens to class I and class II antigens for all patients before HCT; if the PRA shows > 10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained; the donor should be excluded if any of the cytotoxic cross match assays are positive; for those patients with an HLA Class I allele mismatch, flow cytometric or B and T cell cytotoxic cross matches should be obtained regardless of the PRA results; a positive anti-donor cytotoxic crossmatch is an absolute donor exclusion
* DONOR: Patient and donor pairs homozygous at a mismatched allele in the graft rejection vector are considered a two-allele mismatch, i.e., the patient is A*0101 and the donor is A*0102, and this type of mismatch is not allowed
* DONOR: Only filgrastim (G-CSF) mobilized peripheral blood mononuclear cell (PBMC) only will be permitted as a HSC source on this protocol

Exclusion Criteria:

* Patients with rapidly progressive intermediate or high grade NHL
* Patients with a diagnosis of chronic myelomonocytic leukemia (CMML)
* Central nervous system (CNS) involvement with disease refractory to intrathecal chemotherapy
* Presence of circulating leukemic blasts (in the peripheral blood) detected by standard pathology for patients with AML, MDS, ALL or CML
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Females who are pregnant or breast-feeding
* Patients with active non-hematological malignancies (except non-melanoma skin cancers) or those with non-hematological malignancies (except non-melanoma skin cancers) who have been rendered with no evidence of disease, but have a greater than 20% chance of having disease recurrence within 5 years
* Fungal infections with radiological progression after receipt of amphotericin B or active triazole for greater than 1 month
* Cardiac ejection fraction < 35%; ejection fraction is required if age > 50 years or there is a history of anthracycline exposure or history of cardiac disease
* Diffusion capacity of carbon monoxide (DLCO) < 40%, total lung capacity (TLC) < 40%, forced expiratory volume in one second (FEV1) < 40% and/or receiving supplementary continuous oxygen
* The FHCRC PI of the study must approve of enrollment of all patients with pulmonary nodules
* Patients with clinical or laboratory evidence of liver disease would be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension; patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bridging fibrosis, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, or symptomatic biliary disease
* Karnofsky score < 60 or Lansky score < 50
* Patient has poorly controlled hypertension and on multiple antihypertensives
* Human immunodeficiency virus (HIV) positive patients
* Active bacterial or fungal infections unresponsive to medical therapy
* All patients receiving antifungal therapy voriconazole, posaconazole, or fluconazole and who are then randomized to ARM 3 must have rapamycin reduced according to the Standard Practice of Antifungal Therapy Guidelines
* The addition of cytotoxic agents for cytoreduction with the exception of tyrosine kinase inhibitors (such as imatinib), cytokine therapy, hydroxyurea, low dose cytarabine, chlorambucil, or Rituxan will not be allowed within three weeks of the initiation of conditioning
* DONOR: Donor (or centers) who will exclusively donate marrow
* DONOR: Donors who are HIV-positive and/or, medical conditions that would result in increased risk for G-CSF mobilization and harvest of G-PBMC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2004-11; Primary Completion 2011-05 (Actual); Study Completion 2015-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (11):
- United States (7):
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Veterans Administration Center-Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Rigshospitalet University Hospital, Copenhagen, Denmark
- Germany (3):
  - Medizinische Univ Klinik Koln, Cologne
  - Universitaet Leipzig, Leipzig
  - University of Tuebingen-Germany, Tübingen

REFERENCES:
- [Result] Kornblit B, Maloney DG, Storer BE, Maris MB, Vindelov L, Hari P, Langston AA, Pulsipher MA, Bethge WA, Chauncey TR, Lange T, Petersen FB, Hubel K, Woolfrey AE, Flowers ME, Storb R, Sandmaier BM. A randomized phase II trial of tacrolimus, mycophenolate mofetil and sirolimus after non-myeloablative unrelated donor transplantation. Haematologica. 2014 Oct;99(10):1624-31. doi: 10.3324/haematol.2014.108340. Epub 2014 Aug 1. PMID 25085357
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (MMF and Tacrolimus): Patients receive tacrolimus IV or PO every 12 hours on days -3 to 180 with taper beginning on day 100 in the absence of GVHD. Patients also receive Mycophenolate Mofetil [MMF] PO every 8 hours on days 0-29 and then every 12 hours on days 30-96 with taper beginning on day 40 in the absence of GVHD.
  Fludarabine Phosphate: Given IV
  Total-Body Irradiation: Undergo total-body irradiation
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic peripheral blood stem cell transplantation
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic peripheral blood stem cell transplantation
  Tacrolimus: Given IV or PO
  Mycophenolate Mofetil: Given PO
- Arm II (MMF and Tacrolimus Alternate Schedule): Patients receive tacrolimus IV or PO every 12 hours on days -3 to 150 with taper beginning on day 100 in the absence of GVHD. Patients also receive Mycophenolate Mofetil [MMF] PO every 8 hours on days 0-29 and then every 12 hours on days 30-180 with taper beginning on day 150 in the absence of GVHD.
  Fludarabine Phosphate: Given IV
  Total-Body Irradiation: Undergo total-body irradiation
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic peripheral blood stem cell transplantation
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic peripheral blood stem cell transplantation
  Tacrolimus: Given IV or PO
  Mycophenolate Mofetil: Given PO
- Arm III (MMF, Tacrolimus, and Sirolimus): Patients receive tacrolimus and Mycophenolate Mofetil [MMF] as in arm II. Patients also receive sirolimus PO once daily on days -3 to 80.
  Fludarabine Phosphate: Given IV
  Total-Body Irradiation: Undergo total-body irradiation
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic peripheral blood stem cell transplantation
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic peripheral blood stem cell transplantation
  Tacrolimus: Given IV or PO
  Mycophenolate Mofetil: Given PO
  Sirolimus: Given PO
Period: Overall Study
Arm/Group | Arm I (MMF and Tacrolimus) | Arm II (MMF and Tacrolimus Alternate Schedule) | Arm III (MMF, Tacrolimus, and Sirolimus)
Started | 70 | 71 | 69
Completed | 70 | 71 | 69
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (MMF and Tacrolimus) | Arm II (MMF and Tacrolimus Alternate Schedule) | Arm III (MMF, Tacrolimus, and Sirolimus) | Total
Number analyzed (Participants) | 70 | 71 | 69 | 210
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1 | 2
  Between 18 and 65 years | 57 | 50 | 49 | 156
  >=65 years | 13 | 20 | 19 | 52
Age, Continuous [Median (Full Range); unit: years] | 60 [26 to 74] | 60 [13 to 72] | 60 [15 to 75] | 60 [13 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 23 | 82
  Male | 41 | 41 | 46 | 128
Region of Enrollment [Number; unit: participants]
  United States | 59 | 59 | 58 | 176
  Denmark | 5 | 5 | 5 | 15
  Germany | 6 | 7 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grades II-IV Acute GVHD
Description: Number of patients with grades II-IV acute GVHD
  aGVHD Stages
  Skin:
  1. a maculopapular eruption involving < 25% BSA
  2. a maculopapular eruption involving 25 - 50% BSA
  3. generalized erythroderma
  4. generalized erythroderma w/ bullous formation and often w/ desquamation
  Liver:
  1. bilirubin 2.0 - 3.0 mg/100 mL
  2. bilirubin 3 - 5.9 mg/100 mL
  3. bilirubin 6 - 14.9 mg/100 mL
  4. bilirubin > 15 mg/100 mL
  Gut:
  Diarrhea is graded 1 - 4 in severity. Nausea and vomiting and/or anorexia caused by GVHD is assigned as 1 in severity. The severity of gut involvement is assigned to the most severe involvement noted. Patients w/ visible bloody diarrhea are at least stage 2 gut and grade 3 overall.
  aGVHD Grades Grade II: Stage 1 - 2 skin w/ no gut/liver involvement Grade III: Stage 2 - 4 gut involvement and/or stage 2 - 4 liver involvement Grade IV: Pattern and severity of GVHD similar to grade 3 w/ extreme constitutional symptoms or death
Time Frame: 150 days after transplant
Population: Two subjects counted towards accrual but did not proceed to transplant and thus were not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MMF and Tacrolimus) | Arm II (MMF and Tacrolimus Alternate Schedule) | Arm III (MMF, Tacrolimus, and Sirolimus)
Number analyzed (Participants) | 69 | 71 | 68
Participants | 44 | 34 | 32
Statistical Analysis 1: Comparison: Arm I (MMF and Tacrolimus) vs Arm II (MMF and Tacrolimus Alternate Schedule) vs Arm III (MMF, Tacrolimus, and Sirolimus); Test type: Superiority or Other; p = 0.09, Regression, Cox — Overall test of homogeneity among arms, reflecting events over the entire period of follow-up
Statistical Analysis 2: Comparison: Arm I (MMF and Tacrolimus) vs Arm II (MMF and Tacrolimus Alternate Schedule); Test type: Superiority or Other; p = 0.10, Regression, Cox; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.4 to 1.1] — HR for Arm II relative to Arm I, reflecting events over the entire period of follow-u[
Statistical Analysis 3: Comparison: Arm I (MMF and Tacrolimus) vs Arm III (MMF, Tacrolimus, and Sirolimus); Test type: Superiority or Other; p = 0.04, Regression, Cox; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.6 to 1.0] — HR for Arm III relative to Arm I, reflecting events over the entire period of follow-up

2. Secondary Outcome: Number of Non-Relapse Mortalities
Description: Percentage of NRM as estimated by cumulative incidence methods with competing risks.
  Cumulative incidence methods are the standard way to estimate incidence of an endpoint in the presence of competing risks and censoring (ref)" Here is the reference. Gooley TA, Leisenring W, Crowley J, Storer BE: Estimation of failure probabilities in the presence of competing risks: new representations of old estimators. Statistics in Medicine 18:695-706, 1999. PMID 10204198
Time Frame: 200 days after transplant
Population: Two subjects counted towards accrual but did not proceed to transplant and thus were not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MMF and Tacrolimus) | Arm II (MMF and Tacrolimus Alternate Schedule) | Arm III (MMF, Tacrolimus, and Sirolimus)
Number analyzed (Participants) | 69 | 71 | 68
Participants | 3 | 6 | 2
Statistical Analysis 1: Comparison: Arm I (MMF and Tacrolimus) vs Arm II (MMF and Tacrolimus Alternate Schedule) vs Arm III (MMF, Tacrolimus, and Sirolimus); Test type: Superiority or Other; p = 0.55, Regression, Cox — Overall test of homogeneity among arms, reflecting events over the entire period of follow-up

3. Secondary Outcome: Number of Participants Utilizing High-Dose Corticosteroids
Description: Number of patients utilizing high-dose corticosteroids (as a surrogate marker for reduction of acute GVHD), estimated by cumulative incidence methods.
  Cumulative incidence methods are the standard way to estimate incidence of an endpoint in the presence of competing risks and censoring (ref)" Here is the reference. Gooley TA, Leisenring W, Crowley J, Storer BE: Estimation of failure probabilities in the presence of competing risks: new representations of old estimators. Statistics in Medicine 18:695-706, 1999. PMID 10204198
Time Frame: 150 days after transplant
Population: Two subjects counted towards accrual but did not proceed to transplant and thus were not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MMF and Tacrolimus) | Arm II (MMF and Tacrolimus Alternate Schedule) | Arm III (MMF, Tacrolimus, and Sirolimus)
Number analyzed (Participants) | 69 | 71 | 68
Participants | 38 | 35 | 22
Statistical Analysis 1: Comparison: Arm I (MMF and Tacrolimus) vs Arm II (MMF and Tacrolimus Alternate Schedule) vs Arm III (MMF, Tacrolimus, and Sirolimus); Test type: Superiority or Other; p = 0.009, Regression, Cox — Overall test of homogeneity among arms, reflecting events over the entire period of follow-up
Statistical Analysis 2: Comparison: Arm I (MMF and Tacrolimus) vs Arm II (MMF and Tacrolimus Alternate Schedule); Test type: Superiority or Other; p = 0.51, Regression, Cox; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.5 to 1.4] — HR for Arm II relative to Arm I, reflecting events over the entire period of follow-up
Statistical Analysis 3: Comparison: Arm I (MMF and Tacrolimus) vs Arm III (MMF, Tacrolimus, and Sirolimus); Test type: Superiority or Other; p = 0.004, Regression, Cox; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.3 to 0.8] — HR for Arm III relative to Arm I, reflecting events over the entire period of follow-up

4. Secondary Outcome: Number of Participants Surviving Overall
Description: Number of patients surviving, estimated by cumulative incidence methods
  Cumulative incidence methods are the standard way to estimate incidence of an endpoint in the presence of competing risks and censoring (ref)" Here is the reference. Gooley TA, Leisenring W, Crowley J, Storer BE: Estimation of failure probabilities in the presence of competing risks: new representations of old estimators. Statistics in Medicine 18:695-706, 1999. PMID 10204198
Time Frame: 1 Year post-transplant
Population: Two subjects counted towards accrual but did not proceed to transplant and thus were not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MMF and Tacrolimus) | Arm II (MMF and Tacrolimus Alternate Schedule) | Arm III (MMF, Tacrolimus, and Sirolimus)
Number analyzed (Participants) | 69 | 71 | 68
Participants | 48 | 47 | 40
Statistical Analysis 1: Comparison: Arm I (MMF and Tacrolimus) vs Arm II (MMF and Tacrolimus Alternate Schedule) vs Arm III (MMF, Tacrolimus, and Sirolimus); Test type: Superiority or Other; p = 0.93, Regression, Cox — Overall test of homogeneity among arms, reflecting events over the entire period of follow-up

5. Secondary Outcome: Number of Participants Surviving Without Progression
Description: Number of patients with progression-free survival, estimated by cumulative incidence methods
  Cumulative incidence methods are the standard way to estimate incidence of an endpoint in the presence of competing risks and censoring (ref)" Here is the reference. Gooley TA, Leisenring W, Crowley J, Storer BE: Estimation of failure probabilities in the presence of competing risks: new representations of old estimators. Statistics in Medicine 18:695-706, 1999. PMID 10204198
Time Frame: 2 Years post-transplant
Population: Two subjects counted towards accrual but did not proceed to transplant and thus were not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MMF and Tacrolimus) | Arm II (MMF and Tacrolimus Alternate Schedule) | Arm III (MMF, Tacrolimus, and Sirolimus)
Number analyzed (Participants) | 69 | 71 | 68
Participants | 28 | 27 | 26
Statistical Analysis 1: Comparison: Arm I (MMF and Tacrolimus) vs Arm II (MMF and Tacrolimus Alternate Schedule) vs Arm III (MMF, Tacrolimus, and Sirolimus); Test type: Superiority or Other; p = 0.96, Regression, Cox — Overall test of homogeneity among arms, reflecting events over the entire period of follow-up

ADVERSE EVENTS:
Time Frame: AEs: From the start of conditioning to 100 Days post-transplant SAEs: From the start of conditioning to 200 Days post-transplant All-Cause Mortality: Conditioning through 1 Year
Arm/Group | Arm I (MMF and Tacrolimus) | Arm II (MMF and Tacrolimus Alternate Schedule) | Arm III (MMF, Tacrolimus, and Sirolimus)
All-Cause Mortality (participants affected / at risk) | 21/69 | 24/71 | 28/68
Serious Adverse Events (participants affected / at risk) | 9/69 | 8/71 | 7/68
Other Adverse Events (participants affected / at risk) | 25/69 | 22/71 | 25/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (MMF and Tacrolimus) (N=69) | Arm II (MMF and Tacrolimus Alternate Schedule) (N=71) | Arm III (MMF, Tacrolimus, and Sirolimus) (N=68)
Thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Severe hemoptysis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Respiratory infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
CNS cerebrovascular ischemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Toxic leukoencephalopathy, infections w/ pneumonia and pyelonephritis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal pneumatosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GvHD w/ infection (Immune system disorders) | 1 (1) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 1 (1)
Mucormycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GVHD (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (MMF and Tacrolimus) (N=69) | Arm II (MMF and Tacrolimus Alternate Schedule) (N=71) | Arm III (MMF, Tacrolimus, and Sirolimus) (N=68)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 2 (2) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (1) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 4 (4)
Duodenal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 3 (3) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 1 (3) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (9) | 4 (4)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Cervical disk herniation) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Pain, NOS) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Psychosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Pulmonary, NOS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (3)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 2 (3)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Ventricular arrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes